CLINICAL TRIAL: NCT00539084
Title: A Controlled Comparative Pilot Study to Assess the Safety and Efficacy of the MicronJet Microneedle Device Following Intradermal Injection of Lidocaine for Local Anesthesia
Brief Title: A Study to Assess the Safety and Efficacy of a Microneedle Device for Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NanoPass Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP40
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2007-11

CONDITIONS: Local Anesthesia; Intradermal Injections
Keywords: microneedles; microneedle; intradermal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intradermal injection of Lidocaine followed by a painful stimulus (venipuncture)
  Interventions: Device: MicronJet
- 2 (Placebo Comparator): Intradermal injection of placebo followed by a painful stimulus (venipuncture)
  Interventions: Device: MicronJet

INTERVENTIONS:
Device: MicronJet — The MicronJet is a microneedle injection device designed for intradermal delivery of drugs (i.e. delivery into the layers of the skin). In this study the MicronJet will be used to inject Lidocaine or Saline.

SUMMARY:
The purpose of this study is to determine whether the MicronJet microneedle device is effective for inducing rapid and painless local anesthesia prior to insertions of intravenous catheters.

DETAILED DESCRIPTION:
Local anesthesia is routinely administered to reduce patient discomfort and improve the outcome of a wide variety of painful medical procedures. However, injection of a local anesthetic agent into the skin using a regular needle is in itself painful. Therefore, common procedures involving needle pricks (e.g. venipuncture) which may be quite painful are usually performed without local anesthesia.

NanoPass has developed a microneedle injection device (MicronJet) which enables painless delivery of drugs directly into the superficial layers of the skin.

The objective of the study is to assess the safety and efficacy of this device for intradermal injection of a local anesthetic agent before insertion of an intravenous catheter to healthy adults.

Each subject will receive an injection of a local anesthetic to one arm, and a control placebo injection of physiological water to the other arm. Both injections will be administered intradermally using the MicronJet. Following the injections, an intravenous catheter will be inserted into the injection site in each arm, and the subject will rate the pain caused by the insertion. Safety parameters will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females. a signed informed consent.
* No significant abnormalities in screening physical exam.
* No significant abnormalities in clinical laboratory parameters.
* No significant abnormalities in ECG within 21 days of the start of the study.
* Intact skin at the sites of injection.
* Accessible veins in the antecubital area.

Exclusion Criteria:

* Hypersensitivity to local anaesthetics.
* History of previous vasovagal events.
* Presence of tattoos, discoloration, acne, scars, keloids or any other marks, bruises cuts or abrasions at the injection sites.
* Subjects with active or chronic skin disease or systemic disease with significant skin involvement.
* History of skin allergy or hypersensitivity.
* History of easy bruising.
* Current or previous history of neurological disorders (particularly neuropathies).
* A history of drug or alcohol abuse.
* Acute infection within 7 days prior to study day.
* Subjects who participated in a clinical study within 4 weeks prior to study day, or who plan to participate in another clinical trial during the time of the trial.
* Subjects suffering from Behçet's disease.
* Pregnant or lactating women.
* Any contraindication (relative or absolute) to study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Prevalence and intensity of adverse events | 3 Days
Pain scores reported by the subjects following the painful stimulus | one minute after injection

SECONDARY OUTCOMES:
Feedback from study participants and staff on their overall impression with the MicronJet device, using questionnaires | 2 days after injection

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Principal Investigator — Head of the unit for Clinical Research at the Sourasky Medical Center, Tel Aviv, Israel